CLINICAL TRIAL: NCT05894681
Title: Based on the Watson Model for the Prevention of Postpartum Depression Impact of Psychoeducational Intervention
Brief Title: Psychoeducation in Preventing Postpartum Depression According to Watson
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yasemin Ozhuner (Other)
Responsible Party: Sponsor-Investigator, Yasemin Ozhuner, DOCTORATE, Eskisehir Osmangazi University
Organization: Eskisehir Osmangazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YASEMİN ÖZHÜNER
Record Dates: First submitted 2023-02-16; First posted 2023-06-08 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy Related
Keywords: Postpartum depression,; Psychoeducation,; Watson model
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: THE EFFECT OF WATSON MODEL-BASED PSYCOEDUCATIONAL INTERVENTIONS ON PREVENTION OF POSTPARTITION DEPRESS
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): To the intervention group; Training and Care Guide psychoeducation program based on Watson Human Care Theory, prepared for the prevention of postpartum depression, will be implemented as six interviews and each interview will be 90 minutes. Before the psychoeducation, the pregnant women were asked to fill out the Personal Information Form, Edinburgh Postpartum Depression Scale, and the Multidimensional Scale of Perceived Social Support. After the diagnosis with a detailed anamnesis, the Training and Care Guide for the Prevention of Postpartum Depression was applied to the pregnant women with the psychoeducation program and a guide booklet was given to them. The interview was done face to face. Pregnant women were given counseling over the phone when they had questions about education. In the last interview, pregnant women were asked to fill out the Patient Satisfaction Evaluation Form according to Watson Improvement Processes.
  Interventions: Other: THE EFFECT OF WATSON MODEL-BASED PSYCOEDUCATIONAL INTERVENTIONS ON PREVENTION OF POSTPARTITION DEPRESS
- control group (Experimental): Personal Information Form, Edinburgh Postpartum Depression Scale, and Multidimensional Scale of Perceived Social Support were filled in to the control group during the interview. Pregnant women were given routine care applied to pregnant women who applied for antenatal controls in FHCs. The interview was done face to face.
  Interventions: Other: THE EFFECT OF WATSON MODEL-BASED PSYCOEDUCATIONAL INTERVENTIONS ON PREVENTION OF POSTPARTITION DEPRESS

INTERVENTIONS:
Other: THE EFFECT OF WATSON MODEL-BASED PSYCOEDUCATIONAL INTERVENTIONS ON PREVENTION OF POSTPARTITION DEPRESS — THE EFFECT OF WATSON MODEL-BASED PSYCOEDUCATIONAL INTERVENTIONS ON PREVENTION OF POSTPARTITION DEPRESS

SUMMARY:
The postpartum period is marked by significant changes in a woman's priorities, roles, and responsibilities. It is a stressful transition period in which one faces physical and emotional challenges. This stressful transition period. It can seriously affect women's mental health and psychosocial well-being. postpartum depression (PPD) is a common complication in women. PPD in about one in seven women can develop. In addition, PPD is one of the leading causes of maternal morbidity and mortality. Preventive psychosocial and psychological practices are effective in reducing the incidence of PPD. cognitive behavioralist therapy, interpersonal psychotherapy and psychoeducational interventions are among these practices. Counseling, which is traditionally considered as a psychological intervention, is very useful for midwives and nurses. supports a number of theoretical applications and perspectives. Therefore, in order to achieve effective and beneficial results, education should be based on defined and organized theories and models. midwifery and nursing Implementation of care based on a model increases the success of care outcomes. health education Some models in the field allow us to explain the occurrence of behavior and its effect on a particular behavior. Helps us run the health education program to evaluate So about PPD A model selection is necessary for the conceptual framework of knowledge. The model chosen is the change in behavior.

should explain their predictive factors and their effects on PPD. Health education in midwifery and nursing and One of the most frequently used models in the promotion of human care is Watson's Theory of Human Care (IBT). This model is love, It consists of the concepts of compassion, respect, trust and people and is a care that evaluates the individual as a whole provides. When the literature is examined, although there are a few studies aimed at preventing PPD, it is seen that PPD is It has been observed that there is no study on model-based psychoeducational intervention in the prevention of In our study, Watson model applied to pregnant women in the prevention of PPD was used to eliminate this deficiency aimed to evaluate the effect of a psychoeducational intervention based on

DETAILED DESCRIPTION:
The postpartum period is marked by significant changes in a woman's priorities, roles, and responsibilities.

It is a stressful transition period in which physical and emotional difficulties are encountered. This stressful transition period can seriously affect women's mental health and psychosocial well-being.

can affect. Postpartum depression (PPD) is a common complication in women. PPD can develop in approximately one in seven women. In addition, PPD, maternal morbidity and is one of the leading causes of mortality. Preventive psychosocial and psychological practices are effective in reducing the incidence of PPD. Cognitive behavioral therapy, interpersonal psychotherapy, and psychoeducational interventions are among the applications. These interventions have traditionally been face-to-face, individual and group.

format, by phone, online, with peer support, and by trained professionals. can be done. In the meta-analysis results of the randomized controlled trial, psychosocial and psychological interventions It has been found to be effective in preventing PPD. prevalence of PPD 37 randomized and semi-randomized controls evaluated the efficacy of preventive interventions in reducing In this study, it was found that depressive symptoms were significantly lower in the intervention group.

Education given in the perinatal period; mother and family, physical, emotional and mental preparation, health development and by focusing on improved lifestyle behaviors. These trainings are It is of great importance in helping them learn about pregnancy, birth and parenthood. The application of midwifery and nursing care based on a model increases the success of the results. Some models in the field of health education, the formation of behaviors health education program to evaluate our explanation and its impact on a particular behavior.

helps us run. Therefore, a model for the conceptual framework of knowledge about PPD selection is required. The selected model includes the predictive factors of behavioral changes and the impact on PPD.

should explain its effects. Health in midwifery and nursing One of the most frequently used models in education and promotion is Watson's Theory of Human Care (IBT). This The model consists of the concepts of love, compassion, respect, trust and human, and includes the individual as a whole.

provides an evaluative care. Watson's theory suggested that nurses use artistic, encourages the use of aesthetic, spiritual, empirical, political and ethical ways of knowing. their care reach a greater level of awareness of their various physical and non-physical dimensions.

Watson model for nursing practice, 10 important factors in his theory and supports the concept. These factors (10 Healing Processes) are defined as follows:

1. Humanitarian-devotional value system: Adopting values such as humanitarianism and devotion, approach the individual with love and compassion.
2. Instilling faith-hope, honoring the other: Positive health between nurse and patient facilitates promotion.
3. Sensitivity: Developing sensitivity towards oneself and others, through accepting others.

   is the recognition of self-actualization.
4. Help-trust relationship: Developing helping-trusting human care relationship, interpersonal care and is essential for the expression of both positive and negative emotions in the nurse-patient relationship. This is the person effective communication to express emotions and to acknowledge and perceive the emotions of others requires the use of skills.
5. Expression and acceptance of emotions: Encouraging the expression of positive and negative emotions and acceptance is defined as a risk-taking experience for both the patient and the nurse. Nurse and the patient must be prepared for positive or negative feedback.
6. Systematic use of scientific problem solving method in decision making, Scientific contribution to nursing care The nursing process is used to bring a problem-solving approach.
7. Enabling teaching and learning: Promoting interpersonal teaching-learning, care and treatment is an important distinguishing factor. This takes the responsibility from the nurse and puts it on the patient. This concept the nurse to provide the patient with the necessary information and then the responsibility of following up to the patient.

   focus on scrolling.
8. Establishing a suitable environment for recovery: Supportive, protective or corrective mental, physical, Providing the sociocultural and spiritual environment

ELIGIBILITY:
Inclusion Criteria:

* 20-32 weeks of pregnancy,

  * Voluntarily,
  * over 18 years,
  * Literate,
  * Women with a healthy fetus on ultrasonography

Exclusion Criteria:

* • Diagnosed with depression and other mental illness by a physician,

  * Using drugs related to mental illness,
  * Premature birth,
  * Those who did not attend more than one interview

Ages: 20 Weeks to 32 Weeks | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction Evaluation Form According to Watson Improvement Processes | up to the fourth week postpartum
  It is a form developed to evaluate nursing care based on Watson theory. This is a form of satisfaction.
Edinburgh Postpartum Depression Scale | from the 20th week of pregnancy to the fourth postpartum
  Edinburgh Postpartum Depression Scale Edinburgh Postpartum Depression Scale, This scale was used to identify women with postpartum depression
Multidimensional Scale of Perceived Social Support | from the 20th week of pregnancy to the fourth postpartum
  The scale was made to determine the adequacy of social support.
Personal Information Form | up to 32 weeks of pregnancy
  It was prepared to determine the socio-demographic, obstetric history and postpartum depression-related characteristics of the individuals included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Nebahat Özerdoğan, Principal Investigator — Eskisehir Osmangazi University
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chow R, Huang E, Li A, Li S, Fu SY, Son JS, Foster WG. Appraisal of systematic reviews on interventions for postpartum depression: systematic review. BMC Pregnancy Childbirth. 2021 Jan 6;21(1):18. doi: 10.1186/s12884-020-03496-5. PMID 33407226
- [Background] Forster DA, McLachlan HL, Rayner J, Yelland J, Gold L, Rayner S. The early postnatal period: exploring women's views, expectations and experiences of care using focus groups in Victoria, Australia. BMC Pregnancy Childbirth. 2008 Jul 22;8:27. doi: 10.1186/1471-2393-8-27. PMID 18644157
- [Background] Cristescu T, Behrman S, Jones SV, Chouliaras L, Ebmeier KP. Be vigilant for perinatal mental health problems. Practitioner. 2015 Mar;259(1780):19-23, 2-3. PMID 26062269
- [Background] Lau Y, Htun TP, Wong SN, Tam WSW, Klainin-Yobas P. Therapist-Supported Internet-Based Cognitive Behavior Therapy for Stress, Anxiety, and Depressive Symptoms Among Postpartum Women: A Systematic Review and Meta-Analysis. J Med Internet Res. 2017 Apr 28;19(4):e138. doi: 10.2196/jmir.6712. PMID 28455276
- [Background] Dennis CL, Dowswell T. Psychosocial and psychological interventions for preventing postpartum depression. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD001134. doi: 10.1002/14651858.CD001134.pub3. PMID 23450532
- [Background] Sockol LE, Epperson CN, Barber JP. Preventing postpartum depression: a meta-analytic review. Clin Psychol Rev. 2013 Dec;33(8):1205-17. doi: 10.1016/j.cpr.2013.10.004. Epub 2013 Oct 21. PMID 24211712
- [Background] Moshki M, Kharazmi A, Cheravi K, Beydokhti TB. The prediction of postpartum depression: The role of the PRECEDE model and health locus of control. J Family Med Prim Care. 2015 Jul-Sep;4(3):454-60. doi: 10.4103/2249-4863.161354. PMID 26288792
- [Background] Turkel MC, Watson J, Giovannoni J. Caring Science or Science of Caring. Nurs Sci Q. 2018 Jan;31(1):66-71. doi: 10.1177/0894318417741116. PMID 29235958